CLINICAL TRIAL: NCT02964533
Title: Thunder-Fire Moxibustion Therapy for Chronic Fatigue Syndrome on Shenque Acupoint: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Haili Luo, Director, Guangzhou University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20161120
Record Dates: First submitted 2016-11-12; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- TFM (Experimental): thunder-fire moxibustion therapy
  Interventions: Other: thunder-fire moxibustion therapy
- MSM (Active Comparator): common moxa-stick moxibustion therapy
  Interventions: Other: common moxa-stick moxibustion

INTERVENTIONS:
Other: thunder-fire moxibustion therapy — burn moxa stick and heat shenque acupoint
  Arms: TFM
Other: common moxa-stick moxibustion — burn moxa stick and heat shenque acupoint
  Arms: MSM

SUMMARY:
Chronic fatigue syndrome is a group of syndrome and is prevalent in adult. Thunder-fire moxibustion is a commentary therapy belonged to acupuncture therapy. To evaluate the effect and safety of thunder-fire moxibustion therapy for chronic fatigue syndrome, we apply a randomized controlled trial by recruiting chronic fatigue syndrome patient as subject, applying thunder-fire moxibustion on shenque acupoint contrasted to common moxa-stick moxibustion, taking fatigue rating scale score, the content of CD3+、CD4+、CD8+、CD4+/CD8+ as evaluation indexes. The treatment time is 20-30 minutes per session, 3-4 times a week, there are totally 15 sessions.

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinical diagnosis of chronic fatigue syndrome, 2.Age between 18 to 65 years old. 3.Must be able to accept moxibustion treatment 4.Never receive any treatment or has suspended treatment over 2 weeks 5.Patients with good adherence, signed informed consent by themselves

Exclusion Criteria:

* 1.Other primary disease caused by chronic fatigue 2.Pregnancy or breast-feeding women. 3.Merge in other serious diseases, such as severe damage in heart, liver, kidney ,lung or mental illness 4.Has took durg for insomnia treatment 5.Has received acupuncture,massage for chronic fatigue syndrome treatment 6.Suffered from infectious disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
fatigue rating scale score | 5 minutes

SECONDARY OUTCOMES:
content of peripheral t-lymphocyte subsets | 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Haili Luo, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- The Second Clinical Medical College of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Tian L, Wang J, Luo C, Sun R, Zhang X, Yuan B, Du XZ. [Moxibustion at Gaohuang (BL 43) for chronic fatigue syndrome: a randomized controlled trial]. Zhongguo Zhen Jiu. 2015 Nov;35(11):1127-30. Chinese. PMID 26939325